CLINICAL TRIAL: NCT06287138
Title: The Effect of Ciprofol on Breathing Patterns, Respiratory Drive, and Inspiratory Effort in Mechanically Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-182-03
Record Dates: First submitted 2023-12-11; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-12

CONDITIONS: Mechanical Ventilation; Sedation and Analgesia
Keywords: sedation; analgesia; mechanical ventilation; respiratory patterns; respiratory drive; inspiratory effort
MeSH Terms: conditions — Agnosia | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Before the trial drug administration, included patients will receive a continuous infusion of remifentanil for analgesia, starting at 0.01 μg/kg/min and adjusting infusion rate to target a Critical-care Pain Observation Tool (CPOT) score of 0-1. The experimental drug was not to be administered until it was confirmed that the patient's baseline sedation level had reached a RASS score of ≥ -2. For sedation, the ciprofol was started at the rate of 0.3 mg/kg/h and maintained for 30 minutes. Then, the initial infusion rate was increased to 0.4, 0.5, 0.6, 0.7, and up to 0.8 mg/kg/h every 30 minutes. The infusion of ciprofol would be stopped if the RASS score ≤ -4, respiratory rate < 8 breaths/min, or Saturation of pulse oxygen (SpO2) < 90% before the maximal dose of 0.8 mg/kg/h was achieved.
  Interventions: Drug: ciprofol

INTERVENTIONS:
Drug: ciprofol — Ciprofol will be infused at 0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h in sequence for 30 minutes at each dose.

SUMMARY:
Sedatives and analgesics are usually given for analgesic, anxiolytic, or sedating purposes for patients with critical illness, while they inevitably inhibit respiratory and circulatory function. Sometimes, patients receive deep sedation to induce hypoventilation or suppress spontaneous respiratory effort. The sedation level in clinical practice is usually assessed with subjective sedation scoring systems, such as the Richmond Agitation Sedation Scale (RASS). However, studies have found that sedation depth based on RASS is not a reliable marker of respiratory drive during critical illness. In recent years, researchers have proposed to monitor the effects of sedatives and analgesics on respiratory indicators and to implement lung-protective sedation, such as P0.1, Pocc, Pmus, WOB, and PTP. However, different pharmacological characteristics, different depths of sedation, and different sedation regimens among different sedatives and analgesics make a great difference in their effects on respiration. Ciprofol is an analog of propofol, with increased stereoselective effects adding to its anesthetic properties, is increasingly used in the intensive care unit, but its effects on respiration are not well understood. Therefore, this study aims to investigate the effects of ciprofol on respiratory patterns, respiratory drive, and inspiratory effort in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient received surgery under general anesthesia and admitted into the ICU
* The patient has been intubated and is receiving invasively mechanically ventilated with the mode of pressure support (PSV) or continuous positive airway pressure (CPAP)
* The patient requires sedative medication targeting RASS -2 to +1 for comfort, safety and to facilitate the delivery of life support measures

Exclusion Criteria:

* Age < 18 years
* Body mass index (BMI) <18 or >30 kg/m2
* Pregnancy or lactation
* Brain stem tumors, myasthenia gravis, or neuromuscular diseases
* Acute severe neurological disorder and any other condition interfering with RASS assessment
* Systolic blood pressure < 90 mmHg after appropriate intravenous volume replacement and continuous infusions of 2 vasopressors
* Heart rate < 50 beats per minute or second- or third-degree heart block in the absence of a pacemaker
* Contraindicate or allergic to any of the study medications
* Acute hepatitis or serious hepatic dysfunction (Child-Pugh class C)
* Chronic kidney disease with glomerular filtration rate (GFR) < 60 ml/min/1.73m2
* Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Explore the effect of ciprofol on tidal volume | At baseline (before sedation with ciprofol) and 0.3 mg/kg/h ciprofol continuous infusion for 30 minutes
  Change from baseline in tidal volume (ml) at 30 minutes after infusion of ciprofol
Explore the effect of ciprofol on respiratory rate | At baseline (before sedation with ciprofol) and 0.3 mg/kg/h ciprofol continuous infusion for 30 minutes
  Change from baseline in respiratory rate (breaths/min) at 30 minutes after infusion of ciprofol
Explore the effect of ciprofol on minute ventilation | At baseline (before sedation with ciprofol) and 0.3 mg/kg/h ciprofol continuous infusion for 30 minutes
  Change from baseline in minute ventilation (L/min) at 30 minutes after infusion of ciprofol
Explore the effect of ciprofol on P0.1 | At baseline (before sedation with ciprofol) and 0.3 mg/kg/h ciprofol continuous infusion for 30 minutes
  Change from baseline in P0.1 (cmH2O) at 30 minutes after infusion of ciprofol
Explore the effect of ciprofol on PMI | At baseline (before sedation with ciprofol) and 0.3 mg/kg/h ciprofol continuous infusion for 30 minutes
  Change from baseline in PMI (cmH2O) at 30 minutes after infusion of ciprofol
Explore the effect of ciprofol on ΔPocc | At baseline (before sedation with ciprofol) and 0.3 mg/kg/h ciprofol continuous infusion for 30 minutes
  Change from baseline in ΔPocc (cmH2O) at 30 minutes after infusion of ciprofol

SECONDARY OUTCOMES:
Explore the effect of ciprofol on tidal volume | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in tidal volume (ml) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on respiratory rate | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in respiratory rate (breaths/min) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on minute ventilation | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in minute ventilation (L/min) at 30 minutes after infusion of ciprofol at different infusion rates
Explore the effect of ciprofol on P0.1 | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in P0.1 (cmH2O) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on PMI | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in PMI (cmH2O) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on ΔPocc | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in ΔPocc (cmH2O) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on systolic blood pressure | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in systolic blood pressure (mmHg) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on diastolic blood pressure | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in diastolic pressure (mmHg) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on mean arterial pressure | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in mean arterial pressure (mmHg) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on heart rate | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in heart rate (beats/min) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on saturation of pulse oxygen | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in saturation of pulse oxygen (%) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on end-tidal carbon dioxide pressure | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in end-tidal carbon dioxide pressure (mmHg) at 30 minutes after infusion of ciprofol at different rates
Explore the effect of ciprofol on RASS score | At baseline (before sedation with ciprofol) and 30 minutes following each infusion rate adjustment (0.3，0.4，0.5，0.6，0.7，0.8 mg/kg/h)
  Change from baseline in RASS score at 30 minutes after infusion of ciprofol at different rates

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su R, Zhang L, Wang YM, Miao MY, Wang S, Cao Y, Zhou JX. Effects of cipepofol on breathing patterns, respiratory drive, and inspiratory effort in mechanically ventilated patients. Front Med (Lausanne). 2025 Feb 25;12:1539238. doi: 10.3389/fmed.2025.1539238. eCollection 2025. PMID 40070647